CLINICAL TRIAL: NCT02713815
Title: The Repetitive Transcranial Magnetic Stimulation (rTMS) for Amphetamine-type Stimulants Addiction
Brief Title: Novel Intervention for Amphetamine-type Stimulants Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Yunnan Institute For Drug Abuse (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mzhao-004
Record Dates: First submitted 2016-03-07; First posted 2016-03-21 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Amphetamine Addiction
Keywords: Amphetamine-type stimulants; prefrontal-striatal circuits; rTMS; Glutamate/GABA; motivational and cognitive intervention
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Sham Comparator): sham repetitive transcranial magnetic stimulation (rTMS) of the left frontal lobe dorsal lateral effect on ATS dependent induced cognitive dysfunction and other symptoms.
  Interventions: Radiation: sham repetitive transcranial magnetic stimulation (rTMS)
- rTMS group (Active Comparator): Use randomized, prospective pseudo stimulus controlled clinical trial design, evaluation of repetitive transcranial magnetic stimulation of the left frontal lobe dorsal lateral effect on ATS dependent induced cognitive dysfunction and other symptoms.
  Interventions: Radiation: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Radiation: repetitive transcranial magnetic stimulation (rTMS) — Stimulate the dorsomedial prefrontal cortex for 4 weeks by Theta-burst stimulation (TBS), once a day
  Arms: rTMS group
Radiation: sham repetitive transcranial magnetic stimulation (rTMS) — Stimulate the dorsomedial prefrontal cortex for 4 weeks by sham Theta-burst stimulation (TBS), once a day
  Arms: control group

SUMMARY:
The repetitive transcranial magnetic stimulation (rTMS) will be used to treat amphetamine-type stimulant (ATS) addiction.

DETAILED DESCRIPTION:
The Glutamate and GABA deficits in prefrontal cortex play a vital role in ATS addiction and relapse, and proposed repetitive transcranial magnetic stimulation (rTMS) as a novel interventions. Focused on evaluating Glutamate/GABA functions in prefrontal cortex and functional connectivity with deep brain regions, neuropsychological tests, biochemical tests, magnetic resonance spectroscopy (MRS) and functional MRI will be used to investigate the neurobiological mechanism of ATS addiction and relapse. These methods will also be used to evaluate the efficacy of the novel intervention and investigate the mechanisms. The study will be very helpful to develop novel interventions in clinical practice and decrease ATS-related harm for both the patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorders
* Dextromanual

Exclusion Criteria:

* Have a disease that affect cognitive function such as history of head injury, cerebrovascular disease, epilepsy, etc
* Have cognitive-promoting drugs in the last 6 months
* Other substance abuse or dependence in recent five years (except nicotine)
* Mental impairment, Intelligence Quotient (IQ) < 70
* Mental disorders
* Physical disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Craving for ATS assessed by Visual Analog Scales (VAS) at 1 month | Baseline and 1 month
  evaluate all participants' craving for ATS by Visual Analog Scales (VAS)

SECONDARY OUTCOMES:
Number of participants who relapse | 1 month
  Follow up with patients after discharge, evaluate number of participants who relapse
Depression status assessed by Patient Health Questionnaire-9(PHQ-9) | 1 month
  evaluate all participants' depression status by Patient Health Questionnaire-9(PHQ-9)
Anxiety status assessed by Generalized Anxiety Disorder Screener (GAD-7) | 1 month
  evaluate all participants' anxiety status by Generalized Anxiety Disorder Screener (GAD-7)
Cognitive function assessed by Cogstate Battery | 1 month
  evaluate all participants' cognition by Cogstate Battery Chinese version
Functional connectivity assessed by MRI | 1 month
  evaluate all participants' functional connectivity in the brain by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Min, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Gaojing Rehabilitation Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No